CLINICAL TRIAL: NCT03629613
Title: Effects of Oral Antioxidant Cocktail on Vascular Function and Blood Flow in Cardiovascular Disease Patients
Brief Title: Effects of Oral Antioxidant Cocktail in Cardiovascular Disease Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: discontinued due to change in operating plans prior to study initiation and enrollment
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0557-18-FB
Record Dates: First submitted 2018-08-03; First posted 2018-08-14 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — BaseLine dental cement

STUDY DESIGN:
Intervention Model Description: Cardiovascular disease condition; healthy, age-matched control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline (Sham Comparator): Subjects will be tested on one day. Baseline testing will take place and will be followed by oral antioxidant cocktail intake. Oral antioxidant cocktail testing will take place ~2 hours after antioxidant intake.
  During baseline testing, no supplement or placebo intake will be used.
  Interventions: Other: Baseline
- Oral antioxidant cocktail (Experimental): Subjects will be tested on one day. Baseline testing will take place and will be followed by oral antioxidant cocktail intake. Oral antioxidant cocktail testing will take place ~2 hours after antioxidant intake.
  Dose 1:(immediately after baseline) 300 mg alpha-lipoic acid, 500 mg vitamin C, 200 IU vitamin E Dose 2: (30 minutes after dose 1) 300 mg alpha-lipoic acid, 500 mg vitamin C, 400 IU vitamin E
  Interventions: Dietary Supplement: Oral antioxidant cocktail

INTERVENTIONS:
Dietary Supplement: Oral antioxidant cocktail — Oral antioxidant cocktail intake will occur after baseline measurements:
  Dose 1 (immediately after baseline testing): 300 mg alpha-lipoic acid, 500 mg vitamin C, 200 IU vitamin E Dose 2 (30 minutes after Dose 1): 300 mg alpha-lipoic acid, 500 mg vitamin C, 400 IU vitamin E
  Arms: Oral antioxidant cocktail
Other: Baseline — No oral antioxidant cocktail intake or placebo intake will occur prior to baseline measurements
  Arms: Baseline

SUMMARY:
Title: Effects of oral antioxidant cocktail on vascular function and muscle function in cardiovascular disease patients

Cardiovascular disease (CVD) generally refers to various conditions involving narrowed or blocked dysfunctional blood vessels that often lead to heart attack or stroke. One of the main contributors to blood vessel dysfunction is damage to the vascular endothelium. This often results from the accumulation of oxidative stress (OS) and inflammation due to a decrease in blood flow and oxygen transport to the body's organs and skeletal muscle.

The body's natural antioxidant defense system cannot keep up with the high level of OS clearance necessary to maintain proper vascular homeostasis. Previous research has addressed the use of single antioxidants (e.g. vitamin E, beta-carotene, ascorbic acid) in CVD patients, but the use of a combination of antioxidants has yet to be examined. Therefore, the purpose of this study is to examine the effects of acute oral antioxidant cocktail administration (containing vitamin C, E, and alpha-lipoic acid) on oxidative stress, vascular function, autonomic function (heart rate variability), leg blood flow, leg muscle tissue oxygenation, and walking capacity in CVD patients.

This is a parallel study design that will assess the effects of oral antioxidant cocktail administration on CVD patients ages 50-85. Subjects will be required to visit the lab 1 time. This visit will consist of 1) obtaining informed consent and questions, 2) baseline blood sampling and baseline measurements of endothelial function, arterial stiffness, autonomic function (heart rate variability), leg blood flow, leg muscle oxygenation, and a walking test, 3) first dose oral antioxidant cocktail administration followed by a 2-hour break, 4) second dose oral antioxidant cocktail 30 minutes after the first dose, 5) post-consumption blood sampling and measurements of endothelial function, arterial stiffness, autonomic function (heart rate variability), leg blood flow, leg muscle oxygenation, and a walking test.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is one of the leading causes of death in the United States. CVD is attributed to a combination of major risk factors including hypertension, dyslipidemia, obesity, poor diet, low physical activity levels, and vascular endothelial cell dysfunction.

The vascular endothelial cells (VECs) have significant control over vascular homeostatic regulation. In the case of mechanical and chemical stimuli, VECs can release vasoactive substances to regulate vascular tone, cell adhesion, and vascular smooth muscle cell (VSMC) proliferation. When the endothelium is damaged and becomes dysfunctional, atherosclerotic changes take place that can contribute to the development of CVD and atherosclerosis.

Endothelial dysfunction has been partially attributed to high levels of reactive oxygen species (ROS) causing significant oxidative stress (OS). OS is defined as an imbalance between the rate of ROS production and the rate of ROS clearance by the antioxidant defense system, with insufficient clearance leading to oxidative damage of the vasculature. High levels of OS have been shown to negatively affect the vascular endothelium by increasing VSMC proliferation and inflammation, which may result in vascular remodeling. Increased OS also attenuates the bioavailability of nitric oxide, a potent vasodilator, and can further exacerbate the structural and functional changes of the vascular endothelium that are associated with the development of CVD.

When the vascular endothelium becomes dysfunctional (partially due to OS), blood flow and vascular tone regulation become impaired, which then negatively affects O2 transport. Without proper blood flow and O2 transport, exercise capacity becomes attenuated. This is a major concern for CVD patients, because exercise is an effective non-pharmacological therapeutic treatment for many of the CVD risk factors including obesity, dyslipidemia, hypertension, and metabolic syndrome. Therefore, improvement of the antioxidant defense system could alleviate high OS, and improve vasodilatory capacity of blood vessels, blood flow and O2 transport, and by extension, can increase exercise capacity. This would make exercise a more viable treatment option for CVD patients.

The antioxidant defense system contains numerous enzymatic and non-enzymatic antioxidants, including catalase, superoxide dismutase, glutathione peroxidase, vitamins A, E, and C, along with glutathione, ubiquinone, and flavanoids. The antioxidant defense system has been found to be attenuated in CVD patients, particularly in those with peripheral arterial disease. However, as ROS production increases, this antioxidant defense system can be overwhelmed, leading to OS and damage to the tissues. Antioxidant capacity may be improved through supplementation in order to provide better OS clearance in the body, which could then result in better blood flow and O2 delivery to the muscles and other organs in the body.

Previous research has shown that blood flow increases after antioxidant intake. Leg blood flow increased significantly in chronic obstructive pulmonary disease (COPD) patients during knee extension exercise in watts (W) in comparison to healthy age-matched controls (3W: 1,798±128 vs. 1,604±100 mL/min, 6W: 1,992±120 vs. 1,832±109 mL/min, 9W: 2,187±136 vs. 2,035±114 mL/min, P < 0.05, antioxidant supplement vs. control, respectively) following acute antioxidant supplementation (~2 hours prior). In patients with open-angle glaucoma, antioxidant supplementation for one month significantly increased biomarkers of ocular blood flow within the retina and retrobulbar vascular beds, where peak systolic velocity increased by 7.3% (P=0.013) and end diastolic velocity increased by 11% (P=0.014). Cerebral blood flow has also been shown to increase following 12 weeks of antioxidant supplementation. Overall, the use of antioxidant intake, acute and chronic, has shown to improve blood flow to various areas within the vasculature.

Previous research also indicates that the increase in blood flow is indicative of greater O2 supply to the measured area. During knee extension exercise in COPD patients, leg O2 consumption increased significantly in comparison to age-matched controls following acute antioxidant intake (3W: 210±15 vs. 173 ± 12 mL O2/min, 6W: 237±15 vs. 217±14 mL O2/min, 9W: 260±18 mL vs. 244±16 mL O2/min, P< 0.05, antioxidant supplement vs. control, respectively). Following 12 weeks of antioxidant use, oxygen utilization in the right prefrontal cortex increased and was strongly associated with the increase in cerebral blood flow (SO2, from 68.21±1.65% to 66.58±1.58%, P=0.001, pre vs. post, respectively).

Pharmacological interventions are often aimed toward controlling cholesterol and blood pressure; however, OS reduction and vascular endothelial function are not common therapeutic targets. Previous research has addressed the use of antioxidants in CVD patients, but it has focused on the intake of a single antioxidant (e.g. vitamin E, beta-carotene, ascorbic acid) and not a combination of antioxidants. The utilization of a combination of antioxidants and their effects on blood flow and oxygen transport in CVD are as of yet unclear. The purpose of this proposed study is to examine the effects of acute administration of an oral antioxidant cocktail (containing vitamin C, E, and a-lipoic acid E) on oxidative stress, vascular endothelial function, autonomic function, blood flow, and oxygen delivery during a walking test. It is hypothesized that oral antioxidant cocktail administration will reduce oxidative stress markers, and will increase both vascular endothelial function and blood flow, thus increasing oxygen delivery to the muscles and improving walking capacity. This pending data from acute antioxidant administration will give insight to long-term antioxidant use in CVD patients and its effects on oxidative stress, blood flow, and the integration of O2 transport and utilization in the body.

ELIGIBILITY:
Cardiovascular Disease Inclusion Criteria:

1. be able to give written, informed consent
2. be diagnosed with CVD
3. be between 50-85 years old
4. be postmenopausal, meaning having had cessation of menses for at least 12 consecutive months

Healthy Control Inclusion Criteria:

1. be able to give written, informed consent
2. no CVD conditions
3. be between 50-85 years old
4. be postmenopausal, meaning having had cessation of menses for at least 12 consecutive months

Exclusion Criteria (Both Groups):

1. chronic kidney/renal disease
2. chronic heart failure
3. neuromuscular disease
4. known cancer
5. already supplementing with antioxidants or vitamins within 5 days of the study
6. pregnant or nursing women

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Endothelial function | 20 minutes
  Flow-mediated dilation will be used to measure endothelial function in the brachial artery. This will be done pre- and post-antioxidant intake.

SECONDARY OUTCOMES:
Arterial stiffness | 10 minutes
  Brachial-to-ankle pulse-wave velocity and carotid-to-femoral pulse-wave velocity will be used to measure arterial stiffness. This will be done pre- and post-antioxidant intake.
Blood flow | 10 minutes
  Doppler ultrasound will be used to measure blood flow in the femoral and popliteal arteries. This will be done pre- and post-antioxidant intake.
Oxidative stress | 5 minutes
  10 mL of blood will be drawn from an antecubital vein pre- and post-antioxidant intake.
Autonomic function | 40 minutes
  Heart rate variability will be measured to determine autonomic function. This will be done pre- and post-antioxidant intake.
Muscle tissue oxygenation | 28 minutes (during physical walking capacity test)
  Muscle tissue oxygenation will be assessed using near-infrared spectroscopy (NIRS) during a maximal walking protocol pre- and post-antioxidant intake.
Physical walking capacity | 28 minutes
  Physical walking capacity will be measured using the Gardner treadmill protocol pre- and post-antioxidant intake.

CONTACTS AND LOCATIONS:
Overall Officials: Song-Young Park, PhD, Principal Investigator — University of Nebraska

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dahlof B. Cardiovascular disease risk factors: epidemiology and risk assessment. Am J Cardiol. 2010 Jan 4;105(1 Suppl):3A-9A. doi: 10.1016/j.amjcard.2009.10.007. PMID 20102968
- [Background] De Caterina R, Zampolli A, Del Turco S, Madonna R, Massaro M. Nutritional mechanisms that influence cardiovascular disease. Am J Clin Nutr. 2006 Feb;83(2):421S-426S. doi: 10.1093/ajcn/83.2.421S. PMID 16470006
- [Background] Deanfield JE, Halcox JP, Rabelink TJ. Endothelial function and dysfunction: testing and clinical relevance. Circulation. 2007 Mar 13;115(10):1285-95. doi: 10.1161/CIRCULATIONAHA.106.652859. No abstract available. PMID 17353456
- [Background] Ogita H, Liao J. Endothelial function and oxidative stress. Endothelium. 2004 Mar-Apr;11(2):123-32. doi: 10.1080/10623320490482664. PMID 15370071
- [Background] Incalza MA, D'Oria R, Natalicchio A, Perrini S, Laviola L, Giorgino F. Oxidative stress and reactive oxygen species in endothelial dysfunction associated with cardiovascular and metabolic diseases. Vascul Pharmacol. 2018 Jan;100:1-19. doi: 10.1016/j.vph.2017.05.005. Epub 2017 Jun 1. PMID 28579545
- [Background] Szocs K. Endothelial dysfunction and reactive oxygen species production in ischemia/reperfusion and nitrate tolerance. Gen Physiol Biophys. 2004 Sep;23(3):265-95. PMID 15638116
- [Background] Burton GJ, Jauniaux E. Oxidative stress. Best Pract Res Clin Obstet Gynaecol. 2011 Jun;25(3):287-99. doi: 10.1016/j.bpobgyn.2010.10.016. Epub 2010 Dec 3. PMID 21130690
- [Background] Schulz E, Gori T, Munzel T. Oxidative stress and endothelial dysfunction in hypertension. Hypertens Res. 2011 Jun;34(6):665-73. doi: 10.1038/hr.2011.39. Epub 2011 Apr 21. PMID 21512515
- [Background] Trinity JD, Broxterman RM, Richardson RS. Regulation of exercise blood flow: Role of free radicals. Free Radic Biol Med. 2016 Sep;98:90-102. doi: 10.1016/j.freeradbiomed.2016.01.017. Epub 2016 Feb 10. PMID 26876648
- [Background] Poirier P, Despres JP. Exercise in weight management of obesity. Cardiol Clin. 2001 Aug;19(3):459-70. doi: 10.1016/s0733-8651(05)70229-0. PMID 11570117
- [Background] Yoshida H, Ishikawa T, Suto M, Kurosawa H, Hirowatari Y, Ito K, Yanai H, Tada N, Suzuki M. Effects of supervised aerobic exercise training on serum adiponectin and parameters of lipid and glucose metabolism in subjects with moderate dyslipidemia. J Atheroscler Thromb. 2010 Nov 27;17(11):1160-6. doi: 10.5551/jat.4358. Epub 2010 Aug 25. PMID 20805637
- [Background] Hagberg JM, Park JJ, Brown MD. The role of exercise training in the treatment of hypertension: an update. Sports Med. 2000 Sep;30(3):193-206. doi: 10.2165/00007256-200030030-00004. PMID 10999423
- [Background] Tjonna AE, Lee SJ, Rognmo O, Stolen TO, Bye A, Haram PM, Loennechen JP, Al-Share QY, Skogvoll E, Slordahl SA, Kemi OJ, Najjar SM, Wisloff U. Aerobic interval training versus continuous moderate exercise as a treatment for the metabolic syndrome: a pilot study. Circulation. 2008 Jul 22;118(4):346-54. doi: 10.1161/CIRCULATIONAHA.108.772822. Epub 2008 Jul 7. PMID 18606913
- [Background] Urso ML, Clarkson PM. Oxidative stress, exercise, and antioxidant supplementation. Toxicology. 2003 Jul 15;189(1-2):41-54. doi: 10.1016/s0300-483x(03)00151-3. PMID 12821281
- [Background] Pipinos II, Judge AR, Zhu Z, Selsby JT, Swanson SA, Johanning JM, Baxter BT, Lynch TG, Dodd SL. Mitochondrial defects and oxidative damage in patients with peripheral arterial disease. Free Radic Biol Med. 2006 Jul 15;41(2):262-9. doi: 10.1016/j.freeradbiomed.2006.04.003. Epub 2006 Apr 22. PMID 16814106
- [Background] Edwards AT, Blann AD, Suarez-Mendez VJ, Lardi AM, McCollum CN. Systemic responses in patients with intermittent claudication after treadmill exercise. Br J Surg. 1994 Dec;81(12):1738-41. doi: 10.1002/bjs.1800811211. PMID 7827927
- [Background] Frei B. Reactive oxygen species and antioxidant vitamins: mechanisms of action. Am J Med. 1994 Sep 26;97(3A):5S-13S; discussion 22S-28S. doi: 10.1016/0002-9343(94)90292-5. PMID 8085584
- [Background] Rossman MJ, Trinity JD, Garten RS, Ives SJ, Conklin JD, Barrett-O'Keefe Z, Witman MA, Bledsoe AD, Morgan DE, Runnels S, Reese VR, Zhao J, Amann M, Wray DW, Richardson RS. Oral antioxidants improve leg blood flow during exercise in patients with chronic obstructive pulmonary disease. Am J Physiol Heart Circ Physiol. 2015 Sep;309(5):H977-85. doi: 10.1152/ajpheart.00184.2015. Epub 2015 Jul 17. PMID 26188020
- [Background] Harris A, Gross J, Moore N, Do T, Huang A, Gama W, Siesky B. The effects of antioxidants on ocular blood flow in patients with glaucoma. Acta Ophthalmol. 2018 Mar;96(2):e237-e241. doi: 10.1111/aos.13530. Epub 2017 Aug 3. PMID 28772005
- [Background] Nakano M, Murayama Y, Hu L, Ikemoto K, Uetake T, Sakatani K. Effects of Antioxidant Supplements (BioPQQ) on Cerebral Blood Flow and Oxygen Metabolism in the Prefrontal Cortex. Adv Exp Med Biol. 2016;923:215-222. doi: 10.1007/978-3-319-38810-6_29. PMID 27526146
- [Background] Rimm EB, Stampfer MJ, Ascherio A, Giovannucci E, Colditz GA, Willett WC. Vitamin E consumption and the risk of coronary heart disease in men. N Engl J Med. 1993 May 20;328(20):1450-6. doi: 10.1056/NEJM199305203282004. PMID 8479464
- [Background] Klipstein-Grobusch K, den Breeijen JH, Grobbee DE, Boeing H, Hofman A, Witteman JC. Dietary antioxidants and peripheral arterial disease : the Rotterdam Study. Am J Epidemiol. 2001 Jul 15;154(2):145-9. doi: 10.1093/aje/154.2.145. PMID 11447047
- [Background] Ives SJ, Harris RA, Witman MA, Fjeldstad AS, Garten RS, McDaniel J, Wray DW, Richardson RS. Vascular dysfunction and chronic obstructive pulmonary disease: the role of redox balance. Hypertension. 2014 Mar;63(3):459-67. doi: 10.1161/HYPERTENSIONAHA.113.02255. Epub 2013 Dec 9. PMID 24324045
- [Background] Rossman MJ, Groot HJ, Reese V, Zhao J, Amann M, Richardson RS. Oxidative stress and COPD: the effect of oral antioxidants on skeletal muscle fatigue. Med Sci Sports Exerc. 2013 Jul;45(7):1235-43. doi: 10.1249/MSS.0b013e3182846d7e. PMID 23299763